CLINICAL TRIAL: NCT00347672
Title: Phase 1 Inpatient Study of the Safety and Immunogenicity of Live Influenza A Vaccine H5N1 (6-2) AA ca Recombinant (A/VietNam/1203/2004 x A/AnnArbor/6/60/ca), a Live Attenuated Virus Vaccine Candidate for the Prevention of Avian Influenza H5N1 Infection in the Event of a Pandemic
Brief Title: Safety of and Immune Response to a Bird Flu Virus Vaccine (H5N1) in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Johns Hopkins Bloomberg School of Public Health (Other)
Responsible Party: Ruth Karron, MD, Center for Immunization Research (CIR), Johns Hopkins School of Public Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CIR 217; H.22.05.07.22.A2
Record Dates: First submitted 2006-07-03; First posted 2006-07-04 (Estimated); Last update posted 2008-01-21 (Estimated); Status verified 2008-01

CONDITIONS: Influenza; Virus Diseases
Keywords: Bird Flu
MeSH Terms: conditions — Influenza, Human; Virus Diseases; Influenza in Birds

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Two vaccinations of H5N1 VN 2004/AA vaccine at the highest dose
  Interventions: Biological: H5N1 (6-2) AA ca Recombinant (A/VietNam/1203/2004 x A/AnnArbor/6/60/ca)
- 2 (Experimental): One vaccination of H5N1 VN 2004/AA vaccine at a dose in-between the lowest and highest doses
  Interventions: Biological: H5N1 (6-2) AA ca Recombinant (A/VietNam/1203/2004 x A/AnnArbor/6/60/ca)
- 3 (Experimental): One vaccination of H5N1 VN 2004/AA vaccine at the lowest dose
  Interventions: Biological: H5N1 (6-2) AA ca Recombinant (A/VietNam/1203/2004 x A/AnnArbor/6/60/ca)

INTERVENTIONS:
Biological: H5N1 (6-2) AA ca Recombinant (A/VietNam/1203/2004 x A/AnnArbor/6/60/ca) — Live, attenuated recombinant H5N1 (6-2) AA ca Recombinant (A/VietNam/1203/2004 x A/AnnArbor/6/60/ca) vaccine (one of three doses)

SUMMARY:
Avian influenza (AI), or bird flu, has recently become a major health concern in Asia and other parts of the world. The need for a vaccine to prevent the spread of AI among livestock and to humans is sorely needed. The purpose of this study is to test the safety of and immune response to a new AI vaccine in healthy adults.

DETAILED DESCRIPTION:
AI viruses in their natural reservoir in waterfowl are the source from which novel HA and NA subtypes are introduced into the human population, and have the potential to initiate an influenza pandemic. This study will evaluate the safety and immunogenicity of a live, attenuated recombinant AI virus vaccine, H5N1 (6-2) AA Ca Recombinant (A/VietNam/1203/2004 x A/AnnArbor/6/60/Ca).

Participants in this study will receive one or two doses of the vaccine. There are 3 groups in this study:

* Group 1 will receive two vaccinations at the highest dose.
* Group 2 will receive one vaccination at a dose in-between the lowest and highest doses.
* Group 3 will receive one vaccination at the lowest dose.

Group 1 will enroll first, probably in 2006. Groups 2 and 3 will not enroll until it is determined by safety review that the vaccine is well-tolerated and greater than 80% of Group 1 participants shed vaccine virus or develop a specific immune response to the vaccine.

Participation in this study includes a hospital stay in an isolation unit of the Bayview Medical Center of Johns Hopkins University. All participants will receive the vaccine at study entry and will remain in the isolation unit for a minimum of 14 days after vaccination. A physical exam and a nasal wash will occur daily in the isolation unit until a participant is discharged from the hospital. Participants will be allowed to leave the unit once viral cultures for influenza from nasal washes are negative for at least 3 consecutive days beginning on Day 10. Blood collection will occur at study entry, Day 7, sometime between Days 28 and 35, and sometime between Days 56 and 63.

There will be two separate hospitalizations for Group 1 participants. Group 1 participants will receive their doses of vaccine at study entry and sometime between Days 28 and 35. A physical exam and a nasal wash will occur daily in the isolation unit until a participant is discharged from the hospital. Participants will be allowed to leave the unit once viral cultures for influenza from nasal washes are negative for at least 3 consecutive days beginning on Day 10. Blood collection will occur at 4 or 5 selected timepoints, depending on the timing of the second vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Good general health
* Available for the duration of the trial
* Willing to use acceptable forms of contraception

Exclusion Criteria:

* Clinically significant neurologic, cardiac, pulmonary, hepatic, rheumatologic, autoimmune, or renal disease
* Behavioral, cognitive, or psychiatric disease that, in the opinion of the investigator, affects the ability of the volunteer to understand and cooperate with the study
* Medical, work-related, or family problems as a result of alcohol or illicit drug use in the 12 months prior to study entry
* History of severe allergic reaction or anaphylaxis
* Current asthma or reactive airway disease
* History of Guillain-Barre syndrome
* HIV-1 infected
* Hepatitis C virus infected
* Positive for hepatitis B surface antigen (HBsAg)
* Known immunodeficiency syndrome
* Use of corticosteroids or immunosuppressive drugs within 30 days of study entry. Participants who have used topical corticosteroids are not excluded.
* Live vaccine within 4 weeks of study entry
* Killed vaccine within 2 weeks of study entry
* Absence of spleen
* Blood products within 6 months of study entry
* Current smoker
* Have traveled to the Southern Hemisphere or Asia within 14 days prior to study entry
* Have traveled on a cruise ship within 14 days prior to study entry
* Work in the poultry industry
* Investigational agents within 60 days prior to study entry, or currently participating in another investigational vaccine or drug trial
* Allergy to eggs or egg products
* Purified protein derivative (PPD) positive (positive tuberculosis [TB] test)
* Family member with immunodeficiency
* Other condition that, in the opinion of the investigator, would affect the participant's participation in the study
* Pregnant or breastfeeding

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2006-06; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Frequency of vaccine-related reactogenicity events | During the acute monitoring phase of the study
Anti-H5N1 antibody levels and seroconversion, defined as a greater than fourfold rise in serum hemagglutination inhibiting (HI) and/or neutralizing antibody titer compared to Day 0 | Throughout study

SECONDARY OUTCOMES:
To determine the number of vaccinees infected with the H5N1 VN 2004/AA ca recombinant vaccine candidate | Throughout study
If 10^7, 10^5, and 10^3 TCID50 doses of vaccine are administered, to compare the infectivity rates, safety, and immunogenicity between dose groups, and to estimate the HID50 for this vaccine | At study completion
To determine the phenotypic stability of vaccine virus shed | Throughout study
To determine whether immunogenicity is enhanced by a second dose of vaccine, and whether the first dose of vaccine restricts replication of the second dose | Throughout study
To evaluate T-cell mediated and innate immune responses against the H5N1 VN 2004/AA ca recombinant vaccine candidate | Throughout study
To develop a serum bank so that the capacity of the H5N1 VN 2004/AA ca recombinant vaccine candidate to elicit HI and neutralizing antibodies to future H5N1 influenza viruses can be tested | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Ruth A. Karron, MD, Principal Investigator — Center of Immunization Research (CIR), Johns Hopkins Bloomberg School of Public Health
Locations (1):
- Center of Immunization Research (CIR), Johns Hopkins Bloomberg School of Public Health, Baltimore, Maryland, United States

REFERENCES:
- [Background] Ferguson NM, Cummings DA, Cauchemez S, Fraser C, Riley S, Meeyai A, Iamsirithaworn S, Burke DS. Strategies for containing an emerging influenza pandemic in Southeast Asia. Nature. 2005 Sep 8;437(7056):209-14. doi: 10.1038/nature04017. Epub 2005 Aug 3. PMID 16079797
- [Background] Joseph T, Subbarao K. Human infections with avian influenza viruses. Md Med. 2005 Winter;6(1):30-2. PMID 15869106
- [Background] Sims LD, Domenech J, Benigno C, Kahn S, Kamata A, Lubroth J, Martin V, Roeder P. Origin and evolution of highly pathogenic H5N1 avian influenza in Asia. Vet Rec. 2005 Aug 6;157(6):159-64. doi: 10.1136/vr.157.6.159. PMID 16085721
- [Background] Stephenson I, Nicholson KG, Wood JM, Zambon MC, Katz JM. Confronting the avian influenza threat: vaccine development for a potential pandemic. Lancet Infect Dis. 2004 Aug;4(8):499-509. doi: 10.1016/S1473-3099(04)01105-3. PMID 15288823
- [Background] Webby RJ, Perez DR, Coleman JS, Guan Y, Knight JH, Govorkova EA, McClain-Moss LR, Peiris JS, Rehg JE, Tuomanen EI, Webster RG. Responsiveness to a pandemic alert: use of reverse genetics for rapid development of influenza vaccines. Lancet. 2004 Apr 3;363(9415):1099-103. doi: 10.1016/S0140-6736(04)15892-3. PMID 15064027
- [Derived] Karron RA, Talaat K, Luke C, Callahan K, Thumar B, Dilorenzo S, McAuliffe J, Schappell E, Suguitan A, Mills K, Chen G, Lamirande E, Coelingh K, Jin H, Murphy BR, Kemble G, Subbarao K. Evaluation of two live attenuated cold-adapted H5N1 influenza virus vaccines in healthy adults. Vaccine. 2009 Aug 6;27(36):4953-60. doi: 10.1016/j.vaccine.2009.05.099. Epub 2009 Jun 21. PMID 19540952